CLINICAL TRIAL: NCT07162116
Title: A Single-center, Randomized, Double-blind, Placebo- and Positive Drug (Open-label Design) Controlled Phase I Clinical Study to Evaluate the Effect of a Single Oral Dose of XY0206 Tablets on QTc Interval in Healthy Chinese Participants.
Brief Title: A Study to Evaluate the Effect of XY0206 on the QTc Interval in Chinese Healthy Participants
Acronym: XY0206-CQT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: XY0206AML1007
Record Dates: First submitted 2025-08-26; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- XY0206 (Experimental): 12.5 mg/tablet,single dose,administer according to the administration methods of groups A, B, and C.
  Interventions: Drug: XY0206
- Moxifloxacin (Active Comparator): 400mg/tablet,single dose
  Interventions: Drug: Moxifloxacin (400 mg)
- XY0206 Placebo (Placebo Comparator): 12.5 mg/tablet,single dose,administer according to the administration methods of groups A, B, and C.
  Interventions: Other: XY0206 Placebo

INTERVENTIONS:
Drug: XY0206 — 12.5 mg/table,On the morning of the day of dosing , subjects received XY0206 tablets orally on an empty stomach.Each group of 15 subjects was randomly assigned in a 3:1:1 ratio, with 9 receiving XY0206, 3 receiving a placebo of XY0206, and 3 receiving moxifloxacin.Group A (XY0206 tablets: 37.5 mg; moxifloxacin : 400 mg; placebo: 37.5 mg)；Group B(XY0206 tablets: 75 mg; moxifloxacin : 400 mg; placebo: 150mg)；Group C(XY0206 tablets:150 mg; moxifloxacin : 400 mg; placebo: 150mg)
  Arms: XY0206
Drug: Moxifloxacin (400 mg) — 400mg，On the morning of the day of dosing , subjects received moxifloxacin orally on an empty stomach
  Arms: Moxifloxacin
Other: XY0206 Placebo — 12.5mg/table,On the morning of the day of dosing, subjects received XY0206 placebo orally on an empty stomach.Each group of 15 subjects was randomly assigned in a 3:1:1 ratio, with 9 receiving XY0206, 3 receiving a placebo of XY0206, and 3 receiving moxifloxacin.Group A (XY0206 tablets: 37.5 mg; moxifloxacin : 400 mg; placebo: 37.5 mg)；Group B(XY0206 tablets: 75 mg; moxifloxacin : 400 mg; placebo: 150mg)；Group C(XY0206 tablets:150 mg; moxifloxacin : 400 mg; placebo: 150mg)
  Arms: XY0206 Placebo

SUMMARY:
This study plans to enroll 45 (Groups A, B, and C) to 75 healthy participants (including the sample size of other potential dose groups). The participants will be divided into three dose groups: 37.5 mg, 75 mg, and 150 mg. After taking the corresponding investigational product, participants are required to complete test procedures including QTc interval measurement , blood sampling, and vital sign monitoring. The entire test process lasts for 3 days. On the third day, after participants complete laboratory tests and are assessed by physicians as meeting the discharge criteria, they can be discharged.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effect of a single oral dose of XY0206 tablets on the QT/QTc interval in healthy subjects, and to assess the pharmacokinetic (PK) characteristics of XY0206 in healthy humans and its impact on other ECG parameters (HR, PR, QRS interval, T-wave morphology and U-wave presence) in healthy subjects. Additionally, the safety and tolerability of a single oral dose of XY0206 tablets in healthy subjects will be evaluated. Moxifloxacin will be used as a positive control to assess the sensitivity and reliability of this clinical study. This study plans to enroll 45 (Groups A, B, and C) to 75 (including possible additional dose groups) healthy subjects. Group A (XY0206 tablets: 37.5 mg; moxifloxacin hydrochloride tablets: 400 mg; XY0206 placebo: 37.5 mg); Group B (XY0206 tablets: 75 mg; moxifloxacin hydrochloride tablets: 400 mg; XY0206 placebo: 75 mg); Group C (XY0206 tablets: 150 mg; moxifloxacin hydrochloride tablets: 400 mg; XY0206 placebo: 150 mg), with 15 subjects in each group (9 XY0206 tablets, 3 moxifloxacin hydrochloride tablets, and 3 XY0206 placebos). Groups B, C, and possible additional dose groups will follow the "sentinel dosing" approach. Subjects will fast for at least 10 hours the night before dosing. On Day 1, participants will be administered XY0206 tablets, moxifloxacin hydrochloride tablets, or placebo according to the randomization table. XY0206 tablets and placebo will be administered in a double-blind manner, while moxifloxacin hydrochloride tablets will be administered in an open-label manner. Participants will undergo Holter monitoring, PK sample collection, and safety assessment within the specified time frame.

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily sign a written informed consent form.
2. Male or female; aged between 18 and 45 years old (inclusive).
3. Male participants weigh ≥ 50kg, female participants weigh ≥ 45kg, and their body mass index (BMI) is between 19.0 and 26.0 kg/m², inclusive.
4. Physical examination, laboratory tests, and all trial-related examinations (vital signs, electrocardiogram, chest X-ray, abdominal color Doppler ultrasound, etc.) at the screening stage are normal or have only minor abnormalities without clinical significance, and are deemed qualified by the clinical research doctor.
5. Participants can communicate well with the researchers and comply with the protocol requirements to complete the study.

Exclusion Criteria:

Medical history, past medical history, recent medication history:

1. Those with a history of severe systemic diseases (including cardiovascular, digestive, urinary, respiratory systems, etc.), mental disorders, or drug dependence;
2. Those with a history of drug or food allergies, or specific allergies (such as asthma, urticaria, eczema, etc.); or those allergic to XY0206 tablets, moxifloxacin hydrochloride, or other fluoroquinolones, or the excipients contained therein; or those known to be allergic to FLT3 inhibitors;
3. Those with a history of difficulty swallowing or any gastrointestinal diseases (or gastrointestinal resection, etc.) that affect drug absorption;
4. Those with hemorrhoids or perianal diseases with regular/ongoing bleeding, irritable bowel syndrome, inflammatory bowel disease; or those with habitual constipation or diarrhea;
5. Those with a history of pancreatitis;
6. Those who have undergone major surgery within 6 months before screening or whose surgical incisions have not fully healed; major surgeries include but are not limited to any surgeries with significant bleeding risks, prolonged general anesthesia, or incisional biopsies or significant traumatic injuries;
7. Those who have donated blood within 3 months before screening, or plan to donate blood during this study, or have received blood transfusions or lost ≥200ml of blood within 4 weeks before screening;
8. Those who have participated in 4 or more clinical trials within the past year; or those who have participated in any clinical trials and received investigational drugs or devices within 3 months before this trial;
9. Those with a history of drug abuse within the past 5 years or have used drugs within 3 months before the trial;
10. Those who have taken any prescription drugs, over-the-counter drugs, vitamin products, health supplements, or herbal medicines within 4 weeks before screening or within 5 half-lives (if known), whichever is longer; or those who have taken any drugs known to cause QT/QTc interval prolongation or have a risk of causing torsades de pointes (TdP) within 4 weeks before screening;
11. Those with a history of hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia, or hypocalcemia;
12. Those who have received vaccinations within 3 months before screening or plan to receive vaccinations during this study;
13. Those with a history of fainting at the sight of blood or needles and cannot tolerate venous catheterization;

    Health status:
14. Those with neurological, mental, respiratory, cardiovascular, digestive, hematological and lymphatic, endocrine, musculoskeletal, urinary, or any other diseases or physiological conditions that may affect the study results at the time of screening;
15. Those with a history of cardiovascular diseases or risk factors for torsades de pointes (TdP) at the time of screening, including but not limited to: unexplained syncope; heart failure; myocardial infarction; angina pectoris; atrial fibrillation, atrial flutter, atrial premature beats, ventricular premature beats, non-sustained or sustained ventricular tachycardia; bradycardia or sick sinus syndrome; personal or family history of any cardiac conduction abnormalities; long QT syndrome (LQTS) personal or family history; or a family history of sudden death;
16. Those with 12-lead electrocardiogram results exceeding the standard at the screening or baseline period: PR > 200ms, QRS > 110ms, HR < 50 bpm, QTcF > 450 ms (for both males and females); or those with abnormal electrocardiograms and the investigator deems the abnormalities clinically significant (such as atrioventricular block, potential bundle branch block, torsades de pointes (TdP), other types of ventricular tachycardia, ventricular fibrillation and ventricular flutter, clinically significant T-wave changes, or any 12-lead electrocardiogram results that may affect the QTc interval);
17. Those with laboratory test results meeting the following abnormal ranges at the screening or baseline period:

    a. Abnormal hematological indicators: i. White blood cells < lower limit of normal (LLN); ii. Absolute neutrophil count < LLN; iii. Platelet count < LLN; iv. Hemoglobin < LLN. b. Abnormal liver function: AST and/or ALT > upper limit of normal (ULN), total bilirubin and/or direct bilirubin > ULN; c. Creatinine > ULN, creatine kinase > ULN, creatine kinase isoenzyme > ULN, lipase > ULN, amylase > ULN; d. Metabolic abnormalities: serum triglycerides > 1.2 times ULN.
18. Participants with positive hepatitis B surface antigen and/or hepatitis B e antigen, positive hepatitis C antibody, positive human immunodeficiency virus antibody, or positive Treponema pallidum antibody during the screening period;
19. Participants with positive breath alcohol test or positive urine drug abuse screening at baseline;

    Lifestyle restrictions:
20. Participants with special dietary requirements who cannot adhere to the diet and corresponding regulations provided by the clinical research institution;
21. Participants who cannot control special diets (including pitaya, mango, grapefruit and/or xanthine diet, caffeine-containing foods or beverages, strong tea, etc.) during the trial;
22. Participants who have consumed special diets (including pitaya, mango, grapefruit and/or xanthine diet, caffeine-containing foods or beverages, strong tea, etc.) or engaged in vigorous exercise within 48 hours before administration, or have other factors that may affect drug absorption, distribution, metabolism, and excretion;
23. Participants who have consumed alcohol frequently in the 6 months prior to administration, i.e., more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol spirits or 150 mL of wine), or cannot stop alcohol intake during the trial;
24. Participants who smoke more than 5 cigarettes per day in the 3 months prior to administration, or will use any tobacco products during the trial;

    Contraception:
25. Pregnant or lactating women or those with positive pregnancy tests;
26. Participants who have used oral contraceptives within 30 days before screening (applicable to females only);
27. Participants who have used long-acting estrogen or progesterone injections or implants within 6 months before screening (applicable to females only);
28. Females of childbearing age who have had unprotected sexual intercourse with their partners within 14 days before screening;
29. Participants of childbearing age, male or female, who have a plan to conceive from the time of signing the informed consent form until one year after the end of the trial, or who do not agree to use effective contraceptive methods, or do not agree to avoid freezing or donating sperm/eggs.

    Other criteria:
30. Participants who are considered to have poor compliance or have any other factors that make them unsuitable for this trial by the investigator;
31. The investigator, their family members, and related personnel of the research center;
32. Students and subordinates of the investigator, employees of the sponsor, and other vulnerable participants;
33. Participants who may be unable to complete the study for other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
QT/QTc | 48 hours after drug administration
  Holter ECG data of each study participant from 1 hour before administration to 48 hours after administration were collected, and data were extracted according to the collection point to evaluate the effect of a single dose of XY0206 tablets/placebo/moxifloxacin on the QT/QTc interval of healthy people

SECONDARY OUTCOMES:
blood sample | 48 hours after drug administration
  Blood concentration is measured

CONTACTS AND LOCATIONS:
Locations (1):
- PKUCare Luzhong Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: No